CLINICAL TRIAL: NCT05228184
Title: A Randomized Comparative Study Between Liquid (Tirosint®-SOL) and Tablet Formulations of Levothyroxine in Neonates and Infants With Congenital Hypothyroidism
Brief Title: Use of Tirosint®-SOL or Tablet Formulations of Levothyroxine in Pediatric Patients With Congenital Hypothyroidism (CH)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to recruit subjects
Sponsor: IBSA Institut Biochimique SA (Industry)
Collaborators: Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20US-T414
Record Dates: First submitted 2021-12-21; First posted 2022-02-08 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Congenital Hypothyroidism
MeSH Terms: conditions — Congenital Hypothyroidism | interventions — Thyroxine; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Tirosint®-SOL (levothyroxine sodium) oral solution (IBSA Pharma Inc.) at the following strengths: 13, 25, 37.5, 44, 50, 62.5, 75, 88, 100 mcg.
  Interventions: Drug: Tirosint®-SOL
- Control (Active Comparator): Crushed levothyroxine sodium tablets
  Interventions: Drug: Levothyroxine Sodium

INTERVENTIONS:
Drug: Tirosint®-SOL — Dosage will be according to the USPI and Standard of Care.
  Other Names: levothyroxine sodium oral solution (liquid)
  Arms: Treatment
Drug: Levothyroxine Sodium — Tablets will be crushed and dissolved in solution. Dosage will be according to the USPI and Standard of Care.
  Other Names: levothyroxine sodium tablets
  Arms: Control

SUMMARY:
This is a multi-center, prospective, parallel-group, open-label, randomized clinical study in one hundred and twenty-six (126) neonates and infants diagnosed with CH.

Subjects will be randomized in a 2:1 ratio to Treatment (Tirosint®-SOL) or Control (conventional therapy with levothyroxine sodium crushed tablets).

DETAILED DESCRIPTION:
Newly diagnosed neonates will be randomly assigned to start therapy with LT4 at the initial dose recommended by the Standard of Care (SOC). Infants already on LT4 therapy will continue at the same daily dose within the randomly assigned treatment group (dose adjustments are allowed, if needed based on laboratory parameters and clinical response). Once enrolled, subjects will be treated and followed for 12 months (±1.5 months), participating in 7-8 study visits, consisting of 6-7 inclinic and 1-2 (or more if follow-up visits are required) telemedicine (TM) visits. The total number of visits depends on the age at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patient aged 0 to 9 months
* Primary CH diagnosis with elevated TSH and low or normal FT4, requiring treatment with LT4, under either of the following conditions:

  * Neonates newly diagnosed with primary CH and needing to initiate LT4 therapy, or
  * Infants previously diagnosed with primary CH and who are already on LT4 therapy for at least 3 weeks;
* Provide and comply with the informed consent.

Exclusion Criteria:

* Preterm neonates with a gestational age < 37 weeks;
* Low birth weight (LBW) or very low birth weight (VLBW) neonates (weight < 2.5 kg) or VLBW infants (weight < 1.5 kg);
* Neonates in neonatal intensive care units or requiring admission to NICU or neonates/infants hospitalized or requiring hospitalization or in fragile health conditions (e.g. with serious health problems or complications);
* Neonates with CH diagnosis > 4 weeks after delivery;
* Diagnosis of primary gastrointestinal disease:

  * Gastroesophageal reflux requiring medical therapy (beyond thickening of formula or position);
  * Anatomic defects (e.g. intestinal atresia, malrotation, tracheoesophageal fistula, pyloric stenosis, Hirschsprung's disease, gastroschisis);
  * Dietary allergy (e.g. cow's milk protein allergy);
  * Malabsorption related to cystic fibrosis, celiac disease and others;
  * Necrotizing enterocolitis requiring surgical resection;
* Known or suspected adrenal insufficiency (e.g. congenital adrenal hyperplasia, hypopituitarism);
* Diagnosis of congenital cardiac disease, cardiac insufficiency or risk for cardiac failure;
* Diagnosis of chromosomopathy;
* Diagnosis of central hypothyroidism;
* Hypersensitivity to glycerol;
* Concomitant anticonvulsant medications, liothyronine, combination of LT4 and liothyronine, thyroid extracts and/or chronic or long-term use of systemic glucocorticoids
* History of nonadherence with medication or medical visit schedule; or
* Any condition for which, participation would not be in the best interest of the patient or that could limit protocol specified assessments.

Ages: 1 Day to 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
LT4 dose required to maintain TSH in target range (unit: mcg/kg/day) | Up to 22 months based on age group
  The LT4 dose is calculated based on the daily LT4 dose (mcg) used in the time period preceding the visit (or the average daily dose on a weekly basis if more than one strength is used over the course of the week) and the body weight (kg) measured during the visit.

SECONDARY OUTCOMES:
Hormonal profile for TSH | Up to 22 months based on age group
  TSH (unit mU/L)
Hormonal profile for FT4 | Up to 22 months based on age group
  FT4 (unit ng/dL)
Frequency of dose adjustments | Up to 22 months based on age group
  Percent number of subjects (%) who need a dose adjustment in the long-term follow up phase
Number of events of TSH values above 4.5 mU/L | Up to 22 months based on age group
  TSH value above 4.5 mU/L
Number of events of FT4 values below the middle of the laboratory normal range | Up to 22 months based on age group
  FT4 value below the middle of the laboratory normal range
Growth pattern for length of body | Up to 22 months based on age group
  Subject growth measurements in Length (cm) of body
Growth pattern for body weight | Up to 22 months based on age group
  Subject growth measurements in Body weight (kg)
Growth pattern for head circumference | Up to 22 months based on age group
  Subject growth measurements in Head circumference (cm)
Parent/caregiver reports of satisfaction and ease of administration | Up to 22 months based on age group
  Parents Satisfaction Questionnaire is a study-specific tool measuring coping and mental well-being and satisfaction
  Score: 1-Strongly disagree, 2-Disagree, 3-Neutral, 4-Agree, 5-Strongly agree.
Subject acceptance of the treatment (CareCAT) | Up to 22 months based on age group
  Caregiver Administered Children's Acceptance Tool (CareCAT) is a 5-point nominal scale used to assess the acceptance of oral medicines in infants and toddlers who are unable to verbally give their opinion about a medicine
Signs and symptoms of hypothyroidism | Up to 22 months based on age group
  Total number of subjects experiencing hypothyroidism's signs and symptoms
Signs and symptoms of hyperthyroidism | Up to 22 months based on age group
  Total number of subjects experiencing hyperthyroidism's signs and symptoms

OTHER OUTCOMES:
Time to normalize TSH in neonates | Up to 28 days
  Time to normalize TSH into reference range (unit: days)
Time to normalize FT4 in neonates | Up to 28 days
  Time to normalize FT4 into the upper half of the laboratory normal FT4 range (unit: days)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Mautone, Study Director — IBSA Head of R&D Scientific Affairs
Locations (10):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - CHOC Children's Hospital, Orange, California
  - University of California San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Cook Children's Health Care Systems, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No